CLINICAL TRIAL: NCT06728540
Title: Investigation of Physical Activity Levels, Respiratory and Pelvic Floor Muscle Functions of School-Age Children With Lower Urinary Tract Dysfunction
Brief Title: Respiratory and Pelvic Floor Muscle Functions of Children With Lower Urinary Tract Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seda Yakit Yesilyurt (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Seda Yakit Yesilyurt, Assist.prof., Izmir University of Economics
Organization: Izmir University of Economics (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SYY_İEU_3
Record Dates: First submitted 2024-11-06; First posted 2024-12-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Floor Disorders; Lower Urinary Tract Symptoms; Physical Activity
Keywords: Pelvic Floor Disorders,; Lower Urinary Tract Dysfunction; Physical Activity
MeSH Terms: conditions — Pelvic Floor Disorders; Lower Urinary Tract Symptoms; Motor Activity | interventions — Respiratory Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children with Lower Urinary Tract Dysfunction (Study Group) (Experimental): Children included in the study will be evaluated only once. The sociodemographic and clinical characteristics of the children participating in the study will be evaluated with the evaluation form, respiratory muscle strength with the RP Check brand electronic pressure measurement device, and body composition with the Tanita MC-580 brand bioelectrical impedance analyzer. Pelvic floor muscle functions of children with LUTD will be evaluated with the 632 Myomed biofeedback device. The survey questions and the evaluation form will be filled out by the parents.
  Interventions: Other: Investigation of Physical Activity Levels, Respiratory and Pelvic Floor Muscle Function
- Healthy Children (Control Group) (Other): Children included in the study will be evaluated only once. The sociodemographic and clinical characteristics of the children participating in the study will be evaluated with the evaluation form, respiratory muscle strength with the RP Check brand electronic pressure measurement device, and body composition with the Tanita MC-580 brand bioelectrical impedance analyzer. Pelvic floor muscle functions of children with LUTD will be evaluated with the 632 Myomed biofeedback device. The survey questions and the evaluation form will be filled out by the parents.
  Interventions: Other: Investigation of Physical Activity Levels, Respiratory and Pelvic Floor Muscle Function

INTERVENTIONS:
Other: Investigation of Physical Activity Levels, Respiratory and Pelvic Floor Muscle Function — The sociodemographic and clinical characteristics of the children participating in the study will be evaluated with an evaluation form, respiratory muscle strength with an RP Check brand electronic pressure measurement device, and body composition with a Tanita MC-580 brand bioelectrical impedance analyzer. Pelvic floor muscle functions of children with LUTD will be evaluated with a 632 Myomed biofeedback device. The survey questions and the evaluation form will be filled out by the parents.

SUMMARY:
Lower urinary tract dysfunctions (LUTD) are disorders that can occur in the storage and voiding stages of bladder function other than neurological disease or lower urinary tract obstruction. Storage symptoms are increased or decreased voiding frequency, urinary incontinence, urgency and nocturia, while voiding symptoms are classified as hesitation, straining, weak stream and intermittent voiding. Other symptoms are holding maneuvers, feeling of incomplete voiding, post-voiding dripping, genital and lower urinary tract pain. Epidemiological studies show that the prevalence of LUTD is high in school-aged children, with rates as high as 22%. Very little is known about pelvic floor muscle training in children. Relaxation in the pelvic floor muscles is very important for the continuity of micturition and defecation functions. Respiratory function is one of the key elements in the relaxation of the pelvic floor. The relationship of the pelvic floor muscles with the diaphragm and their role in intra-abdominal pressure regulation have been demonstrated by many studies. In the adult population, it has been emphasized that the respiratory pattern should be corrected in pelvic floor dysfunctions and pelvic floor muscle training should be provided in those with respiratory problems. In the literature, rehabilitation programs for children with LUTD are treatment approaches in which respiratory and pelvic floor muscle training are applied together, but it has not been clearly stated which isolated approach is responsible for the resulting effect. In addition, these studies have emphasized that diaphragmatic exercises reduce or improve symptoms through the relaxation mechanism they create in the abdominal wall. However, unlike the literature, one of the aims of this study is to reveal the relationship between inspiratory and expiratory muscle strength and LUTD.

ELIGIBILITY:
Inclusion Criteria in LUTD group:

* Diagnosed with LUTD,
* Nighttime enuresis at least twice a week for at least 3 consecutive months.
* Daytime enuresis at least once a month for at least 3 consecutive months.
* Girls aged 6-14,
* who consent to participate in the study with the consent of their mother and father or legal guardian (legal representative) will be included in the study.

Inclusion Criteria for healthy individuals in the study:

* Girls aged 6-14,
* who consent to participate in the study with the consent of their mother and father or legal guardian (legal representative) will be included in the study.

Exclusion Criteria:

* Children under 6 years of age,
* Anatomical changes in the urinary system,
* Spina bifida,
* History of active urinary tract infection,
* Neurological disease,
* An accompanying respiratory system disease (asthma and a history of frequent upper respiratory tract infections),
* Cognitive impairment,
* Mental retardation,
* Chronic kidney disease,
* Who have previously undergone orthopedic surgery will not be included in the study.

Ages: 6 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Strength of Respiratory Muscle | baseline
  To measure respiratory muscle strength, maximal inspiratory pressure (MIP or PImax) and maximal expiratory pressure (MEP or PEmax) measurements will be used with a non-invasive, RP Check brand electronic pressure measuring device.
Level of Physical Activity | baseline
  Physical Activity Questionnaire for Children (PAQ-C):The physical activity levels of children will be assessed using the Physical Activity Questionnaire for Children (PAQ-C). The PAQ-C was developed in Canada to evaluate moderate to vigorous physical activity levels. It is based on the child's self-reported recall of the previous 7 days. The PAQ-C consists of 10 items, with 9 items used to calculate the activity score.
  The first question includes a list of 22 commonly performed activities. Responses to this question are evaluated on a 5-point scale (1 = never, 5 = 7 times or more). An average score is calculated, with higher scores indicating higher levels of physical activity.

SECONDARY OUTCOMES:
Voiding Disorders | baseline
  Voiding Disorders Symptom Score (VOS):The severity of voiding dysfunction symptoms in children will be assessed using the Voiding Dysfunction Symptom Score. This score was developed by Akbal et al. in 2005 and consists of 14 questions in total. Thirteen of the questions evaluate symptoms related to daytime urinary incontinence, nighttime urinary incontinence, daily voiding frequency, the presence of constipation, and various symptoms associated with urinary incontinence. The 14th question assesses the impact of these symptoms on quality of life. The total score of the scale ranges from 0 to 35 points, with higher scores indicating increased severity of voiding dysfunction symptoms.
Bladder and Bowel Dysfunction | baseline
  Bladder and Bowel Dysfunction Scale (BDS):The severity of children's bladder and bowel dysfunction symptoms will be assessed with the Bladder and Bowel Dysfunction Scale. The MBDS was developed by Afshar et al. in 2009. Bladder and bowel dysfunction symptoms are assessed and diagnosed with this scale. Its Turkish validity and reliability were made by Kaya Narter et al. in 2017. The scale consists of 14 questions. The first 13 questions are specific to bladder and bowel dysfunction symptoms. The last question questions the degree of difficulty of completing the survey. Each question is a 5-point Likert type and the last question is not added to the scoring. The total score varies between 0-52 and an increase in the score means an increase in symptom severity.
Functions of Pelvic Floor Muscle | baseline
  After a brief informative training using visuals about pelvic floor muscles and their functions, the electrical activity of the pelvic floor muscles of children with LUTD will be measured with the 632 Myomed biofeedback device.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No